CLINICAL TRIAL: NCT03326258
Title: Phase Ib/II Clinical Trial of Glembatumumab Vedotin and Nivolumab in Advanced Solid Tumors
Brief Title: Glembatumumab Vedotin, Nivolumab, and Ipilimumab in Treating Patients With Advanced Metastatic Solid Tumors That Cannot Be Removed by Surgery
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study itself was Disapproved on 04/20/2018 and will not be moving forward.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01979; NCI-2017-01979 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10157 (Other: Duke University - Duke Cancer Institute LAO); 10157 (Other: CTEP); UM1CA186704 (NIH)
Record Dates: First submitted 2017-10-30; First posted 2017-10-31 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-05

CONDITIONS: Advanced Malignant Solid Neoplasm; Estrogen Receptor Negative; GPNMB Positive; HER2/Neu Negative; Metastatic Malignant Solid Neoplasm; Metastatic Melanoma; Progesterone Receptor Negative; Stage III Breast Cancer AJCC v7; Stage III Cutaneous Melanoma AJCC v7; Stage III Uveal Melanoma AJCC v7; Stage IIIA Cutaneous Melanoma AJCC v7; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Breast Cancer AJCC v6 and v7; Stage IV Cutaneous Melanoma AJCC v6 and v7; Stage IV Uveal Melanoma AJCC v7; Triple-Negative Breast Carcinoma; Unresectable Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma; Breast Neoplasms; Uveal Melanoma; Triple Negative Breast Neoplasms | interventions — glembatumumab vedotin; CR011-vcMMAE; Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (glembatumumab vedotin, nivolumab, ipilimumab) (Experimental): Patients receive glembatumumab vedotin IV over 90 minutes and nivolumab IV over 60 minutes on day 8 of course 1 and on day 1 of subsequent courses. Patients in melanoma expanded cohort also receive ipilimumab IV over 90 minutes on day 1. Treatment with ipilimumab repeats every 21 days for 4 courses in the absence of disease progression or unaccepted toxicity and courses with glembatumumab vedotin and nivolumab repeat every 21 days in the absence of disease progression or unaccepted toxicity.
  Interventions: Drug: Glembatumumab Vedotin; Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Other: Pharmacological Study

INTERVENTIONS:
Drug: Glembatumumab Vedotin — Given IV
  Other Names: Antibody-Drug Conjugate CR011-vcMMAE; CDX-011; CR011-vcMMAE; CR011-vcMMAE Immunotoxin
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase Ib/II trial studies the best dose of glembatumumab vedotin when giving together with nivolumab and ipilimumab in treating patients with solid tumor that has spread to other places in the body and cannot be removed by surgery. Monoclonal antibodies, such as glembatumumab vedotin, nivolumab, and ipilimumab, may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase 2 dose (RP2D) for the combination of glembatumumab vedotin and nivolumab in patients with solid tumors. (Phase Ib) II. To evaluate the antitumor activity of the combination in 4 expansion cohorts (melanoma, uveal melanoma, GPNMB overexpressing triple negative breast cancer [TNBC], other GPNMB overexpressing solid tumors) as measured by overall response by Immune-Modified Response Evaluation Criteria in Solid Tumors (iRECIST)/Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. (Phase II)

SECONDARY OBJECTIVES:

I. To characterize the safety and toxicity profile of the combination. II. To evaluate the clinical benefit rate (no disease progression within 6 months), progression free survival (PFS), and overall survival (OS) in patients receiving the combination treatment.

III. To evaluate the pharmacokinetics (PK) of glembatumumab vedotin and nivolumab in combination in serum and in mononuclear phagocyte system (MPS) cells in peripheral blood mononuclear cells.

IV. Profile differences in the type, number and density of Fc-receptors (FcgammaR) on MPS cells in blood of patients prior to and after administration of glembatumumab vedotin and nivolumab as a method to evaluate the factors affecting PK and pharmacodynamics (PD) variability and mechanisms of drug-drug interactions.

V. Characterize differences in chemokines (CCL2 and CCL5) and other cytokines in blood of patients prior to and after administration of glembatumumab vedotin and nivolumab as a method to evaluate the factors affecting PK and PD variability and mechanisms of drug-drug interactions.

VI. To evaluate the pharmacodynamic (PD) effects of the combination in plasma and tissue biomarkers.

OUTLINE:

Patients receive glembatumumab vedotin intravenously (IV) over 90 minutes and nivolumab IV over 60 minutes on day 8 of course 1 and on day 1 of subsequent courses. Patients in melanoma expanded cohort also receive ipilimumab IV over 90 minutes on day 1. Treatment with ipilimumab repeats every 21 days for 4 courses in the absence of disease progression or unaccepted toxicity and courses with glembatumumab vedotin and nivolumab repeat every 21 days in the absence of disease progression or unaccepted toxicity.

After completion of study treatment, patients are followed up for 4 weeks and then at 30 and 70 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative measures do not exist or are no longer effective
* For TNBC and solid tumors other than melanoma: GPNMB expression as defined by at least 25% of malignant epithelial cells or tumor stromal cells expression GPNMB at any intensity via central immunohistochemistry on archived or biopsied tumor tissue (as per standard clinical care) from an advanced/metastatic disease site; for melanoma or uveal melanoma cohort: GPNMB testing results will not be required for eligibility assessment
* Patients must have measurable disease, in addition to at least one lesion in a reasonably safe location for study-related biopsies; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) by chest x-ray or as >= 10 mm (>= 1 cm) with computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Willing to undergo study-related biopsies as noted in study calendar: before treatment, after glembatumumab-only, and after combination therapy
* Prior treatment with immune checkpoint inhibitors or antibody drug conjugates are allowed.

  * For cutaneous melanoma cohort, patients should have received PD-1/CTLA-4 targeting therapy in combination and had disease progression
  * For all other cohorts including phase Ib dose-finding, patients should have received at least one line of standard non-immunotherapy treatment
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 80%)
* Life expectancy of greater than 12 weeks
* Leukocytes >= 2,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 75,000/mcL
* Hemoglobin >= 9.0 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (except patients with Gilbert syndrome, who can have total bilirubin < 3.0 mg/dL)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional upper limit of normal (or =< 5.0 x institutional upper limit of normal in presence of metastatic liver disease)
* Serum creatinine =< 1.5 x institutional upper limit of normal OR creatinine clearance >= 50 mL/min (if using the Cockcroft-Gault formula)
* Women of childbearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; WOCBP should use an adequate method to avoid pregnancy for 32 weeks after the last dose of investigational drug; women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of nivolumab; women must not be breastfeeding; men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year; men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product; women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile as well as azoospermic men) do not require contraception; women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal; menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes; in addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she (or the participating partner) should inform the treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had systemic therapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) or radiotherapy within 2 weeks prior to entering the study
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities >= grade 2 other than alopecia)
* Patients who are receiving any other concurrent investigational agents; those with history of receiving investigational cancer treatment are allowed as long as washout period is fulfilled
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression; patients with treated and stable brain metastases will be allowed; controlled brain metastases are defined as no radiographic progression for at least 4 weeks following radiation and/or surgical treatment (or 4 weeks of observation if no intervention is clinically indicated), and off of steroids for at least 2 weeks, and no new or progressive neurological signs and symptoms
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab, glembatumumab vedotin, or other agents used in study; this includes sensitivity to the drugs dolastatin or auristatin
* History of severe hypersensitivity reaction to any monoclonal antibody
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Participants must not have a history of life-threatening toxicity related to prior IO treatment (eg, anti-CTLA-4 or anti-PD-1/PD-L1 treatment or any other antibody or treatment specifically targeting T-cell co-stimulation or immune checkpoint pathways); i) participants with toxicities that are unlikely to recur with standard countermeasures (eg, hormone replacement treatment after adrenal crisis) are eligible
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with nivolumab and glembatumumab vedotin
* Human immunodeficiency virus (HIV) patients should be allowed if otherwise eligible, with the following caveats:

  * Undetectable HIV viral load by standard clinical assay
  * Willing to remain adherent with antiretroviral therapy that has minimal overlapping toxicity or pharmacokinetic interactions with protocol therapy
  * CD4+ T cell counts of 200/mm^3 or greater
  * No acquired immunodeficiency syndrome (AIDS)-defining events other within the past 12 months
  * Near normal life expectancy if not for presence of the cancer
  * Not taking antiviral agents that are otherwise prohibited because of CYP interactions
* Patients should be excluded if they have a positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded; these include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease; patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible; patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible
* Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses =< 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease; patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption); physiologic replacement doses of systemic corticosteroids are permitted, even if =< 10 mg/day prednisone equivalents; a brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* Patients who have had evidence of active or acute diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation should be evaluated for the potential need for additional treatment before coming on study
* Use of any vaccines against infectious diseases (e.g. influenza, varicella, pneumococcus) within 4 weeks of initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Recommended phase 2 dose for the combination of glembatumumab vedotin and nivolumab (Phase Ib) | Up to 21 days
  All adverse events and toxicities will be tabulated and reported by type and grade for all dose levels of all treatment combinations and the proportions will be reported with exact 90% binomial confidence intervals.
Antitumor activity measured by Immune-Modified Response Evaluation Criteria in Solid Tumors (iRECIST)/Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (Phase II) | Up to 70 days
  Descriptive statistics and graphical analysis will be used to summarize patients' demographic and clinicopathological characteristics, patient safety and efficacy outcomes and correlative markers. Overall response rates will be calculated and 2-sided 90% confidence intervals will also be provided for each cohort.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 70 days
  Will be assessed by Common Terminology Criteria for Adverse Events version 4.03. Will be tabulated and reported by type and grade for each cohort and the proportions will be reported with exact 90% binomial confidence intervals.
Overall response rate | Up to 70 days
  Will be analyzed by the Kaplan-Meier method. The association between subgroups of interest and response to treatment will be assessed using Fisher's exact test.
Clinical benefit rate | Up to 70 days
  Will be analyzed by the Kaplan-Meier method. The association between subgroups of interest and response to treatment will be assessed using Fisher's exact test.
Progression free survival | Up to 70 days
  Will be analyzed by the Kaplan-Meier method. The association between subgroups of interest and response to treatment will be assessed using Fisher's exact test.
Overall survival | Up to 70 days
  Will be analyzed by the Kaplan-Meier method. The association between subgroups of interest and response to treatment will be assessed using Fisher's exact test.
Pharmacokinetic parameters | Up to 70 days
  The pharmacokinetics (PK) of glembatumumab vedotin and nivolumab in combination in serum and in mononuclear phagocyte system (MPS) cells in peripheral blood mononuclear cells will also be assessed descriptively. The descriptive statistics of plasma concentration-time data will first be tabulated. PK parameters will be estimated using both standard non-compartmental and compartmental methods. A repeated measurement statistical model will also be used to perform intra patient evaluation of changes in PK.
Levels of plasma and tissue biomarkers | Up to 70 days
  PD-L1 and other immune biomarkers including tumor infiltrating lymphocytes before and after treatment (after glembatumumab vedotin, and then after the combination) will be described using summary statistics. The change of immune markers will be assessed using linear mixed model for repeated measurement data. Data transformation will be performed if necessary to better satisfy the assumption of normality distribution. Univariate and multivariate logistic regression models will be used to evaluate predictive ability of these baseline biomarkers on the response to the combination of glembatumumab vedotin and nivolumab. Receiver operating characteristic (ROC) curves will be used to explore the optimal cut-off points for each biomarker to differentiate responders versus non-responders. The predictive ability will also be summarized using the area under ROC curves (AUC), and the 95% confidence intervals of AUC will be obtained using bootstrap resampling methods.

CONTACTS AND LOCATIONS:
Overall Officials: Haeseong Park, Principal Investigator — Duke University - Duke Cancer Institute LAO